CLINICAL TRIAL: NCT06008106
Title: Efficacy and Safety of Tunlametinib Capsules Versus Combination Chemotherapy of Investigator's Choice in Advanced NRAS-mutant Melanoma Patients Who Had Previously Received Immunotherapy
Brief Title: Comparing Tunlametinib Capsules and Combination Chemotherapy in Advanced NRAS-mutant Melanoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Kechow Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL-085-301
Record Dates: First submitted 2023-08-08; First posted 2023-08-23 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Melanoma
Keywords: Mitogen-Activated Protein Kinase Kinases; NRAS; Melanoma
MeSH Terms: conditions — Melanoma | interventions — CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tunlametinib (Experimental): Drug tunlametinib will be administered as 12mg BID
  Interventions: Drug: tunlametinib
- Assigned Interventions (Active Comparator): combination chemotherapy
  Interventions: Drug: paclitaxel +carboplatin, or temozolomide +cisplatin, or dacarbazine +cisplatin

INTERVENTIONS:
Drug: tunlametinib — 12mg BID
  Arms: tunlametinib
Drug: paclitaxel +carboplatin, or temozolomide +cisplatin, or dacarbazine +cisplatin — according to investigators' suggestion
  Arms: Assigned Interventions

SUMMARY:
This is a multicenter, two-arm, open-label, randomized controlled phase III clinical trial to evaluate the efficacy and safety of tunlametinib capsule in comparison with the combination chemotherapy of investigator's choice in advanced melanoma patients with NRAS mutation who have received immunotherapy before. Subjects were stratified according to the baseline lactate dehydrogenase level and chemotherapy.

DETAILED DESCRIPTION:
A total of 165 subjects will be included and randomly assigned to the corresponding treatment group in a 2:1 ratio by Interactive Web Response System（IWRS）.

Experimental group: subjects received continuous administration of tunlametinib capsules every 28 days, and the study treatment was terminated until intolerable toxicity, disease progression, withdrawal of informed consent, death, or when the risk outweigh the benefit assessed by the investigators, or when the study was terminated (whichever occurred earlier).

Control group: subjects received the combination chemotherapy (paclitaxel +carboplatin, or temozolomide +cisplatin, or dacarbazine +cisplatin, investigator's choice according to the conditions of the subjects) every 28 days until intolerable toxicity, disease progression, withdrawal of informed consent, death, or when the risk outweigh the benefit assessed by the investigator or when the study was terminated (whichever occurred earlier).

Efficacy was evaluated by independent radiology review committee and the investigator, respectively.

Within 30 days after the last administration of the study drug, the safety of the subjects will also be closely monitored and recorded. After safety visit or the last administration of the study drug (whichever occurs later), subject survival follow-up is conducted every 12 weeks to confirm the survival status and record new anti-tumor treatment until death, lost to follow-up, withdrawal of informed consent, or the end of this study (whichever occurs earlier).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Patients with unresectable stage III or metastatic IV melanoma confirmed by histology or cytology.
3. History of immunotherapy failure or could not tolerate immunotherapy
4. NRAS mutation at baseline;.
5. There is at least one lesion that can be evaluated as target lesions according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
6. Eastern cooperative oncology group (ECOG) performance status of grade 0-1.
7. Life expectancy > 3 months.
8. No major surgery (excluding baseline tumor biopsy) or major trauma occurred at least 4weeks prior to investigational drug administration.
9. Left ventricular ejection fraction (LVEF) ≥ 50% within 7 days before dosing according to echocardiographic findings.
10. Key laboratory tests must be conducted within 7 days before dosing and meet the inclusion criteria:
11. Able to understand and voluntarily sign the Informed Consent Form.
12. Patients must be willing and able to complete the study procedure and follow-up examination.

Exclusion Criteria:

* Exclusion Criteria:

  1. Having the following treatment before receiving the study drug: ① received chemotherapy, targeted therapy or other study drug treatment within 4 weeks before the first administration or within 5 half lives of the drug (whichever is longer); ② received immunotherapy and biological therapy within 4 weeks before the first administration; ③ received traditional Chinese medicines with anti-tumor activities approved by National Medical Products Administration (NMPA) within 2 weeks before the first administration.;
  2. The toxic reactions of previous anti-tumor treatment have not been recovered;
  3. Current use of other anti-cancer drugs.
  4. Subjects with symptomatic or untreated brain metastasis, meningeal metastasis or spinal cord compression except for subjects with asymptomatic brain metastasis;
  5. History of any of the following within 6 months of screening: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass grafting, symptomatic congestive heart failure, severe heart arrhythmia requiring medication, uncontrolled hypertension, cerebrovascular accident, or transient ischemic attack, diabetic ketoacidosis, deep vein thrombosis, or symptomatic pulmonary embolism.
  6. ECG Corrected Q-T interval formula (QTcB) ≥ 480 msec (adjusted by Bazett's formula) during screening, or a history of congenital long QT syndrome.
  7. History or current evidence of retinal diseases;
  8. Previous or current neuromuscular diseases related to CK elevation;
  9. Previous or current interstitial lung disease or interstitial pneumonitis;
  10. Uncontrolled concomitant diseases or infectious diseases.
  11. Bleeding symptoms of grade 3 as defined by the National Cancer Institute General Terminology Standard for Adverse Events (NCI CTCAE V5.0) within the 4 weeks prior to study initiation.
  12. Inability to swallow the capsule, refractory nausea and vomiting, malabsorption, external biliary diversion, or any small intestinal resection that would preclude adequate absorption of the study drug.
  13. Patients who are receiving and cannot discontinue regimen-prohibited intravenous or oral drugs that affect CYP isoenzymes (strong inducers and strong inhibitors of CYP2C9) at least 1 week prior to initiation of study treatment and during the study period.
  14. Patients with a history of malignancy within the past 5 years;
  15. Human immunodeficiency virus (HIV) antibody positive; syphilis antibody (anti-TP) positive; Hepatitis C virus (HCV) antibody positive and HCV RNA positive; HBsAg positive and HBV DNA positive.
  16. Patients who have been previously treated with MEK inhibitors.
  17. Patients with known hypersensitivity to investigational drug, proposed chemotherapy or their analogues.
  18. History of allogeneic bone marrow transplantation or organ transplantation.
  19. Serum pregnancy test results are positive for premenopausal female patients;
  20. Other severe, acute, or chronic clinical or psychiatric disorders or laboratory abnormalities that may increase the risk and interfere with the study results in the opinion of investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2027-09-22 (Estimated); Study Completion 2027-09-22 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival(PFS) | up to 12 months
  defined as the time from first dose to the earliest documented disease progression or death due to any cause

SECONDARY OUTCOMES:
Overall survival(OS) | up to 12 months
  defined as the time from the date of taking drugs to the date of death due to any cause
Duration of response(DOR) | up to 12 months
  Duration of response is defined as subjects who show a confirmed clinical response (CR) or partial response (PR), the time from first documented evidence of CR or PR until the first documented sign of disease progression or death
Disease control rate(DCR) | up to 12 months
  Proportion of subjects with response defined as CR, PR, and SD throughout the study from subjects first dose to disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Hongqi Tian, phD, Study Director — Shanghai Kechow Pharma, Inc.
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No